CLINICAL TRIAL: NCT00995384
Title: A Novel Modality of Cardiac CT in Characterization of Acute Infective Endocarditis
Brief Title: Cardiac Computed Tomography (CT) Scan Compared to Transesophageal Echocardiogram (TEE) in Endocarditis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HIC 2009-148; R/C# 98699; RI-09-17
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2012-03

CONDITIONS: Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT scan (Other): CT Scan for endocarditis patients. All patients receive intervention.
  Interventions: Procedure: CT Scan

INTERVENTIONS:
Procedure: CT Scan — Cardiac CT with special attention to valves in Endocarditis patients.

SUMMARY:
The purpose of this study is to assess the effectiveness of cardiac CT versus TEE in endocarditis patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute endocarditis with positive TEE

Exclusion Criteria:

* Renal failure
* Contrast dye allergy
* Beta-blocker allergy

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Visual Difference in CT versus TEE images in Endocarditis | Upon CT Scan

SECONDARY OUTCOMES:
Morbidity | 4 weeks & 6 months post CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Kadaj, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hosptial, Royal Oak, Michigan, United States